CLINICAL TRIAL: NCT06925243
Title: Neoadjuvant Apatinib Combined With Sintilimab and Perioperative SOX Versus Neoadjuvant Sintilimab Combined With Perioperative SOX for Intestinal Type of Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma: A Prospective, Multicenter, Open-Label, Randomized Controlled Phase III Study
Brief Title: Neoadjuvant Apatinib Combined With Sintilimab and Perioperative SOX Versus Neoadjuvant Sintilimab Combined With Perioperative SOX for Intestinal Type of Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zuoyi Jiao (Other)
Responsible Party: Sponsor-Investigator, Zuoyi Jiao, Medical Professor, Lanzhou University Second Hospital
Organization: Lanzhou University Second Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LanzhouU2H-2025A-120
Record Dates: First submitted 2025-03-30; First posted 2025-04-13 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Gastric Cancer (Including Stomach and Gastroesophageal Junction [GEJ]); Neoadjuvant Therapy; Adjuvant Chemotherapy; pCR Rate; MPR; ORR,OS,PFS
Keywords: apatinib; sintilimab; SOX; Neoadjuvant therapy; gastric cancer; intestinal type
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant apatinib combined with sintilimab and perioperative SOX group (Experimental): Participants will receive an intravenous injection of sintilimab (200 mg) combined with the SOX regimen (oxaliplatin 130 mg/m² and S-1, with the initial dose determined based on body surface area). Additionally, apatinib (250 mg) will be administered orally once daily during the first three neoadjuvant cycles. This treatment will be administered for three to four cycles prior to surgery, followed by radical surgery, including D2 or D2+ lymph node dissection. Within 3 to 6 weeks post-surgery, patients will begin adjuvant SOX chemotherapy. Postoperative patients will receive four cycles of adjuvant SOX chemotherapy, administered every three weeks.
  Interventions: Drug: Neoadjuvant apatinib combined with sintilimab and perioperative SOX
- Neoadjuvant sintilimab combined with perioperative SOX group (Active Comparator): Participants will receive an intravenous injection of sintilimab (200 mg) combined with the SOX regimen (oxaliplatin 130 mg/m² and S-1, with the initial dose determined based on body surface area). This treatment will be administered for three to four cycles prior to surgery, followed by radical surgery, including D2 or D2+ lymph node dissection. Within 3 to 6 weeks post-surgery, patients will begin adjuvant SOX chemotherapy. Postoperative patients will receive four cycles of adjuvant SOX chemotherapy, administered every three weeks.
  Interventions: Drug: Neoadjuvant sintilimab combined with perioperative SOX

INTERVENTIONS:
Drug: Neoadjuvant apatinib combined with sintilimab and perioperative SOX — Sintilimab: 200mg, iv, day 1 Oxaliplatin: 130 mg/m², iv, day 1 S-1: 40-60 mg/m², po, day 1-14 (BSA < 1.25 m², 40 mg bid, 1.25 m² ≤ BSA < 1.5 m², 50 mg bid, BSA ≥ 1.5 m², 60 mg bid) Apatinib: 250mg, po, day1-21, for 3 cycles preoperatively
  Arms: Neoadjuvant apatinib combined with sintilimab and perioperative SOX group
Drug: Neoadjuvant sintilimab combined with perioperative SOX — Sintilimab: 200mg, iv, day 1 Oxaliplatin: 130 mg/m², iv, day 1 S-1: 40-60 mg/m², po, day 1-14 (BSA < 1.25 m², 40 mg bid, 1.25 m² ≤ BSA < 1.5 m², 50 mg bid, BSA ≥ 1.5 m², 60 mg bid)
  Arms: Neoadjuvant sintilimab combined with perioperative SOX group

SUMMARY:
This study aims to compare the efficacy and safety of neoadjuvant apatinib combined with sintilimab and perioperative SOX chemotherapy versus neoadjuvant sintilimab combined with perioperative SOX chemotherapy in locally advanced intestinal-type gastric cancer/gastroesophageal junction adenocarcinoma. The primary questions include:

1. Whether the complete remission rate (pCR) of the apatinib combined with sintilimab and SOX regimen is higher than that of the sintilimab combined with SOX regimen.
2. The safety of the apatinib combined with sintilimab and SOX regimen.

Participants will be divided into:

1. Experimental Group: Participants will receive an intravenous injection of sintilimab (200 mg) combined with the SOX regimen (oxaliplatin 130 mg/m² and S-1, with the initial dose determined based on body surface area). Additionally, apatinib (250 mg) will be administered orally once daily during the first three neoadjuvant cycles.
2. Control Group: Participants will receive treatment with the sintilimab combined with the SOX regimen.

This treatment will be administered for three to four cycles prior to surgery, followed by radical surgery, including D2 or D2+ lymph node dissection. Surgery is scheduled four weeks after the last neoadjuvant therapy (NAT) cycle. Within 3 to 6 weeks post-surgery, patients will begin adjuvant SOX chemotherapy. Postoperative patients will receive four cycles of adjuvant SOX chemotherapy, administered every three weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Type of Participant and Disease Characteristics

   1. Patients must have a pathologically confirmed diagnosis of HER-2 negative tumor and intestinal type gastric or gastroesophageal junction adenocarcinoma according to Lauren's histological subtypes.
   2. Patients must have previously untreated locally advanced gastric or gastroesophageal junction adenocarcinoma (stage cT2 to cT4), with lymph nodes ranging from N0 to N3 and no evidence of metastatic disease (M0).
   3. Patients with Siewert type 2 or 3 tumors are eligible. Enrollment of participants with Siewert type 1 tumors will be limited to those for whom the planned treatment is perioperative chemotherapy and resection.
2. Demographics

   1. Male or female subjects must be between the ages of ≥ 18 and ≤ 75 years at the time of signing the informed consent.
   2. Expected Survival: The expected survival time must be ≥ 12 weeks.
   3. Performance Status: Subjects must have an ECOG performance status of 0 or 1.
   4. Male Contraception: Non-sterilized male subjects who are sexually active with a female partner of childbearing potential must use an effective method of contraception from Day 1 through 120 days after receipt of the final dose of the investigational product. It is strongly recommended for the female partner of a male subject to also use an effective method of contraception throughout this period.
   5. Female subjects of childbearing potential must be willing to use adequate contraception methods throughout the study and for 120 days after the last dose of the study drug. The decision to discontinue contraception after this time point should be discussed with the attending physician. Periodic abstinence, contraceptive rhythm methods, and withdrawal are not acceptable forms of contraception.

      * Females of childbearing potential are defined as those who are not surgically sterile (e.g., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause).
      * Highly effective contraception methods, resulting in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, are required. Acceptable methods include a combination of a hormonal method (e.g., contraceptive pill) and a barrier method (e.g., male condom plus spermicide) to prevent pregnancy.
      * Barrier methods include male condom plus spermicide, copper T intrauterine device, and levonorgestrel-releasing intrauterine system.

   ii.Hormonal methods include implants, hormone injection, combined pill, minipill, and patch.
   * If a female subject becomes pregnant or suspects pregnancy during her participation in the study or her partner's participation, she must promptly inform her treating physician.
3. Organ Function

   1. Blood Routine (no blood transfusion within 14 days): WBC ≥ 3.0 × 10^9/L; ANC ≥ 1.5 × 10^9/L; PLT ≥ 100 × 10^9/L; HGB ≥ 80 g/L.
   2. Hepatic Function: Total bilirubin (TBIL) ≤ 1.5 × ULN, or direct bilirubin ≤ ULN for those with total bilirubin levels 1.5 × ULN and ALT/AST levels ≤ 2.5 × ULN.
   3. Renal Function: Creatinine (Cr) ≤ 1.5 × ULN or Creatinine Clearance (CrCl) ≥ 60 mL/min for those with Cr > 1.5 × ULN.
   4. Coagulation Function: INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN.
   5. Cardiac Function: Cardiac function will be assessed using electrocardiogram and color Doppler ultrasound, and subjects must have had no myocardial infarction within the last six months. Hypertension and other coronary heart diseases must be controllable.

      * Females of childbearing potential are defined as those who are not surgically sterile (e.g., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause).
      * Highly effective contraception methods, resulting in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, are required. Acceptable methods include a combination of a hormonal method (e.g., contraceptive pill) and a barrier method (e.g., male condom plus spermicide) to prevent pregnancy.
      * Barrier methods include male condom plus spermicide, copper T intrauterine device, and levonorgestrel-releasing intrauterine system.

   iv.Hormonal methods include implants, hormone injection, combined pill, minipill, and patch.
   * If a female subject becomes pregnant or suspects pregnancy during her participation in the study or her partner's participation, she must promptly inform her treating physician.
4. Informed Consent All subjects must provide written informed consent to participate in the study.
5. Other Inclusions

   1. Prior Treatment: Patients must not have previously received any anti-tumor treatments, including radiotherapy, chemotherapy, targeted therapy, or immunotherapy.
   2. Plan to proceed to surgery following pre-operative chemotherapy based on standard staging studies per local practice.

Be willing to provide tissue and blood sample from a tumor lesion at baseline and at time of surgery

Exclusion Criteria:

1. Medical Conditions

   1. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
   2. Has a known additional malignancy that is progressing or has required active treatment within the past 5 years (except for cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, or carcinoma in situ that has undergone potentially curative therapy).
   3. Has an active infection requiring systemic therapy.
   4. Has an active autoimmune disease that has required systemic treatment in the past 2 years. (NOTE: Subjects with vitiligo, alopecia, Grave's disease, Type I diabetes mellitus, hypothyroidism (e.g., following Hashimoto's syndrome) only requiring hormone replacement on a stable dose (without adjustment in the first 4 weeks of study treatment), psoriasis or eczema not requiring systemic treatment (within the past 2 years), or conditions not expected to recur in the absence of an external trigger are not excluded.)
   5. Has any complications requiring systemic treatment with corticosteroids such as prednisone (> 10mg/day) or other immunosuppressive medications within 14 days prior to the first administration. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is allowed.
   6. History of primary immunodeficiency.
   7. Has received a live vaccine or other immune-activating anti-tumor drugs (such as interferon, interleukin, thymosin, or immunotherapy) within 30 days prior to the first dose of study treatment.
   8. Has a known history of active tuberculosis.
   9. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
   10. Has a known severe allergy or hypersensitivity to sintilimab or apatinib or any of the study chemotherapy agents and/or to any of their excipients.
   11. Presence of any of the following cardiovascular and cerebrovascular diseases or cardiovascular and cerebrovascular risk factors:

       * Grade II or higher myocardial ischemia or myocardial infarction, poorly controlled arrhythmia (including QTc interval ≥ 480 ms), grade III or IV cardiac insufficiency, or left ventricular ejection fraction (LVEF) < 50.0% as determined by ultrasonic cardiography.
       * Cerebrovascular accident, transient ischemic attack, or other arteriovenous thrombotic, embolic, or ischemic events.
2. Prior/Concomitant Therapy

   1. Subjects who have already enrolled in another clinical study, unless it is an observational, non-interventional clinical study, or they are in the follow-up period for an interventional study.
   2. Subjects who have received any systemic or curative anti-tumor therapy, including radiotherapy, chemotherapy, targeted therapy.
   3. Subjects who have previously received any anti-PD-1, anti-PD-L1 antibody, or any other antibody or drug therapy targeting T-cell co-stimulation or checkpoint pathway, e.g. ICOS or agonists (e.g., CD40, CD137, GITR, and OX40, etc.).
3. Other exclusion criteria

   1. Confirmed HER-2 positive tumor will be excluded.
   2. Patients could not provide tumor samples and blood samples.
   3. Pregnant or lactating patients, as well as patients with childbearing potential who plan to be pregnant within 5 months after the study; Women of childbearing should receive a blood pregnancy test within 7 days before the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Enrollment to surgical treatment takes about 4 months.
  Pathological Complete Response rate (pCR) refers to the proportion of cases in which no active cancer cells are detected in the surgically resected tumor tissue after neoadjuvant therapy, as assessed using the Becker TRG grading system.

SECONDARY OUTCOMES:
Major pathological response (MPR) rate | Enrollment to surgical treatment takes about 4 months.
  Major Pathological Response (MPR) rate refers to the proportion of patients who, after receiving neoadjuvant therapy, are assessed using the Becker TRG grading system and have less than 10% residual viable cancer cells in the surgically resected tumor tissue.
Objective response rate (ORR) | From enrollment to preoperative imaging assessment, it takes approximately 4 months.
  The Objective Response Rate (ORR) is a widely used efficacy measure in clinical trials, especially in oncology, to assess the objective changes in tumors in response to treatment. It represents the proportion of patients whose tumors have achieved either a Complete Response (CR) or a Partial Response (PR). The assessment of ORR is typically based on the internationally standardized criteria for evaluating solid tumor responses, known as RECIST v1.1 (Response Evaluation Criteria in Solid Tumors, version 1.1).
3-year survival rate (3-year OS rate) | From the point of enrollment to the end of the 3-year follow-up period.
  The 3-year survival rate (3-year OS rate) is the percentage of patients who survive 3 years after enrollment.
Adverse Event | From enrollment to the completion or discontinuation of treatment, an estimated duration of eight months is expected.
  For the classification and grading of Adverse Events (AEs), the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 is generally used as the standard.
Disease control rate (DCR) | From enrollment to preoperative imaging assessment, it takes approximately 4 months.
  DCR is the percentage of patients with measurable disease at baseline who experience CR, PR, or SD, as determined by BICR using RECIST v1.1 guidelines.
3-year event-free survival rate (3-year EFS rate). | From the point of enrollment to the end of the 3-year follow-up period.
  3-year EFS rate is defined as the proportion of patients who remain free from disease recurrence, progression, or death over a three-year period, without experiencing any predefined adverse events.
R0 resection rate | Enrollment to surgical treatment takes about 4 months.
  The R0 resection rate is defined as the proportion of patients in whom no cancer cells are detected at the surgical margins under microscopic examination, indicating complete removal of the tumor with no visible residual cancer, both macroscopically and microscopically.
Downstaging rates of T, N, TNM stages. | Enrollment to preoperative imaging assessment takes about 4 months.
  The tumor downstage rate represents the percentage of patients whose overall ypTNM, T, or N stage has decreased from their baseline cTNM, cT, or cN stage. Tumor staging was assessed using baseline cTNM and postoperative ypTNM evaluations according to the 8th edition of the AJCC Gastric Cancer Staging Manual.
Surgery-related complications | Enrollment to surgical treatment takes about 4 months.
  Surgery-related complications are defined as any complications occurring within 30 days following surgery, classified according to the Clavien-Dindo Classification of Surgical Complications. These complications include, but are not limited to, vomiting, fever, incision infection, post-operative pneumonia, anastomotic hemorrhage or leakage, chylous leakage, pneumonia, intestinal obstruction, and other related issues.
Programmed death-ligand 1 combined positive score (PD-L1 CPS) | After enrollment, the measurements were completed.
  PD-L1 expression acts as a predictive biomarker for assessing treatment efficacy, encompassing metrics such as the pathologic complete response rate (pCR rate), major pathologic response rate (MPR rate), and both the 3-year overall survival rate (OS rate) and 3-year Event-Free Survival (EFS) rate.
Microsatellite instability (MSI) status | After enrollment, the measurements were completed.
  Microsatellite instability status acts as a predictive biomarker for assessing treatment efficacy, encompassing metrics such as the pathologic complete response rate (pCR rate), major pathologic response rate (MPR rate), and both the 3-year overall survival rate (OS rate) and 3-year Event-Free Survival (EFS) rate.
The ratio of NG2+/CD31 | Enrollment to surgical treatment takes about 4 months.
  The ratio of NG2+/CD31 acts as a predictive biomarker for assessing treatment efficacy, encompassing metrics such as the pathologic complete response rate (pCR rate), major pathologic response rate (MPR rate), and both the 3-year overall survival rate (OS rate) and 3-year Event-Free Survival (EFS) rate.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - First Hospital of Lanzhou University, Lanzhou, Gansu
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The Gastrointestinal Surgery Department, Sun Yat-sen University Cancer Center Gansu Hospital, Lanzhou, Gansu

IPD SHARING:
Plan to Share IPD: No